CLINICAL TRIAL: NCT02197806
Title: Safety and Efficacy of AGN-199201 and AGN-190584 in Patients With Presbyopia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 199201-007
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-10

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AGN-199201 (Experimental): 1 drop of AGN-199201 ophthalmic solution followed by 1 drop of AGN-199201 vehicle in the non-dominant eye and 2 drops of AGN-199201 vehicle in the dominant eye, once and twice daily for 3 days each.
  Interventions: Drug: AGN-199201; Drug: AGN-199201 Vehicle
- AGN-190584 (Experimental): 1 drop of AGN-190584 ophthalmic solution followed by 1 drop of AGN-199201 vehicle in the non-dominant eye and 2 drops of AGN-199201 vehicle in the dominant eye, once and twice daily for 3 days each.
  Interventions: Drug: AGN-190584; Drug: AGN-199201 Vehicle
- AGN-199201 + AGN-190584 in One Eye (Experimental): 1 drop of AGN-199201 ophthalmic solution followed by 1 drop of AGN-190584 ophthalmic solution in the non-dominant eye and 2 drops of AGN-199201 vehicle in the dominant eye, once and twice daily for 3 days each.
  Interventions: Drug: AGN-199201; Drug: AGN-190584; Drug: AGN-199201 Vehicle
- AGN-199201 + AGN-190584 in Both Eyes (Experimental): 1 drop of AGN-199201 ophthalmic solution followed by 1 drop of AGN-190584 ophthalmic solution in both eyes, once and twice daily for 3 days each.
  Interventions: Drug: AGN-199201; Drug: AGN-190584

INTERVENTIONS:
Drug: AGN-199201 — 1 to 2 drops of AGN-199201 ophthalmic solution in the eye(s) as per protocol.
  Arms: AGN-199201; AGN-199201 + AGN-190584 in Both Eyes; AGN-199201 + AGN-190584 in One Eye
Drug: AGN-190584 — 1 to 2 drops of AGN-190584 ophthalmic solution in the eye(s) as per protocol.
  Arms: AGN-190584; AGN-199201 + AGN-190584 in Both Eyes; AGN-199201 + AGN-190584 in One Eye
Drug: AGN-199201 Vehicle — 1 to 2 drops of AGN-199201 vehicle in the eye(s) as per protocol.
  Arms: AGN-190584; AGN-199201; AGN-199201 + AGN-190584 in One Eye

SUMMARY:
A study to evaluate the safety and efficacy of AGN-199201 alone, AGN-190584 alone and concurrent use of AGN-199201 and AGN-190584 in patients with presbyopia (inability to focus for near vision).

ELIGIBILITY:
Inclusion Criteria:

-Presbyopia in each eye that impacts daily activities.

Exclusion Criteria:

* Use of any topical ophthalmic medications, including artificial tears
* Contact lens use in either eye within 14 days or planned use during the study
* History of eye surgery
* Diagnosis of any type of glaucoma or ocular hypertension

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Newport Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AGN-199201 | AGN-190584 | AGN-199201 + AGN-190584 in One Eye | AGN-199201 + AGN-190584 in Both Eyes
Started | 15 | 17 | 16 | 17
Completed | 15 | 16 | 16 | 16
Not Completed | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN-199201 | AGN-190584 | AGN-199201 + AGN-190584 in One Eye | AGN-199201 + AGN-190584 in Both Eyes | Total
Number analyzed (Participants) | 15 | 17 | 16 | 17 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.9 (3.88) | 49.1 (3.47) | 48.7 (4.16) | 49.1 (3.97) | 49.2 (3.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 7 | 10 | 43
  Male | 2 | 4 | 9 | 7 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least a 2 Line Improvement From Baseline in Uncorrected Near Visual Acuity (UNVA) in the Non-Dominant Eye
Description: UNVA is assessed without corrective lenses in the non-dominant eye. UNVA is measured using an eye chart and is reported as the number of lines read correctly. The lower the number of lines read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of lines read correctly means that vision has improved. The percentages of patients with at least a 2 or more line improvement in UNVA in the non-dominant eye are presented.
Time Frame: Baseline, Day 3
Population: Modified Intent to Treat: all randomized patients with a baseline assessment and at least 1 postbaseline assessment of UNVA
Measure: Number; unit: Percentage of Patients
Arm/Group | AGN-199201 | AGN-190584 | AGN-199201 + AGN-190584 in One Eye | AGN-199201 + AGN-190584 in Both Eyes
Number analyzed (Participants) | 15 | 17 | 16 | 16
Percentage of Patients | 46.7 | 70.6 | 56.3 | 68.8

ADVERSE EVENTS:
Description: The Safety Population included all patients who received at least 1 dose of study treatment and was used to assess adverse events (AEs) and serious adverse events (SAEs).
Arm/Group | AGN-199201 | AGN-190584 | AGN-199201 + AGN-190584 in One Eye | AGN-199201 + AGN-190584 in Both Eyes
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17 | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 5/15 | 4/17 | 8/16 | 5/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AGN-199201 (N=15) | AGN-190584 (N=17) | AGN-199201 + AGN-190584 in One Eye (N=16) | AGN-199201 + AGN-190584 in Both Eyes (N=17)
Vision Blurred (Eye disorders) | 0 | 1 | 2 | 1
Conjunctival Hyperaemia (Eye disorders) | 0 | 1 | 1 | 1
Lacrimation Increased (Eye disorders) | 0 | 1 | 1 | 1
Metamorphopsia (Eye disorders) | 0 | 0 | 0 | 1
Ocular Discomfort (Eye disorders) | 0 | 0 | 2 | 0
Eyelid Retraction (Eye disorders) | 4 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0
Eye Irritation (Eye disorders) | 0 | 1 | 0 | 0
Punctate Keratitis (Eye disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Product Taste Abnormal (General disorders) | 0 | 0 | 0 | 1
Discomfort (General disorders) | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.